CLINICAL TRIAL: NCT06905574
Title: Postoperative Analgesic Efficacy of Intraoperative Surgeon-Guided Serratus Block: A Prospective Randomized Study
Brief Title: Surgeon-Guided Serratus Block in Breast Reduction Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: alperen can kokten (Other)
Responsible Party: Sponsor-Investigator, alperen can kokten, doctor faculty member, Samsun University
Organization: Samsun University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: SGSB-01; SamsunU (Other: Samsun university)
Record Dates: First submitted 2025-02-10; First posted 2025-04-01 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Postoperative Pain Control; Breast Reduction
Keywords: breast reduction; postoperative pain control

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Control (No Intervention): No intervention will be made in this group.
- Group SSPB (Experimental): Surgeon guided serratus block will be applied before closing dermoglandular flaps
  Interventions: Other: surgeon guided serratus block

INTERVENTIONS:
Other: surgeon guided serratus block — Surgeon guided Serratus Block will be applied before closing dermoglandular flaps
  Arms: Group SSPB

SUMMARY:
Surgeon guided serratus block, which can be performed by the surgeon in participants undergoing breast reduction surgery, may reduce the sensation of pain from the surgical field in the postoperative period. Thus, participants experience less pain in the postoperative period, consume less analgesics, and there is a decrease in related complications. The aim of this study was to evaluate the effects of the intraoperative surgeon guided serratus block applied on the analgesic consumption of the participants in the first 24 hours after surgery in participants undergoing breast reduction surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patient's willingness to be included in the study
* 18-65 years
* Woman
* Operated with inferior pedicled breast reduction technique
* The distance from the sternal notch to the nipple complex is between 25-40cm
* ASA I-II
* Breast Usg result BIRADS 1-2
* Patients who have not previously received RT to the breast and have no history of malignancy

Exclusion Criteria:

* Patient's request/refusal not to be included in the study
* Previous history of malignancy
* RT story,
* ASA 3-4-5-patient group
* Severe organ failure
* Alcohol, drug addiction
* Bupivacaine allergy
* Diagnosis of psychiatric illness and psychiatric drug use
* Surgery lasting longer than 3 hours
* Bleeding diathesis

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 60 (Actual)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-10-30 (Actual); Study Completion 2025-10-31 (Actual)

PRIMARY OUTCOMES:
24 hours postoperatively opioid consumption | 24 hours
  In the postoperative period, patients will be given opioids according to their pain density with a patient-controlled device, and the daily Morphine consumption in Patient Controlled Analgesia device will be collected and compared between groups.

SECONDARY OUTCOMES:
post-operative acute pain status, post-operative nausea-vomiting status, post-operative NRS determination of pain at rest and in motion determination of complications such as nausea, vomiting, itching, determination of the first PCA analgesic request. | 24 hours
  Changes in the Numerical Rating Scale (NRS) will be recorded at rest and during movement. The participant's baseline NRS will be recorded, followed by measurements before and after neuraxial positioning and up to 24 hours post-surgery. The NRS is a unidimensional measure of pain intensity in adults. The 11-point numerical scale ranges from '0' representing one end of the pain spectrum (e.g. 'no pain') to '10' representing the other end (e.g. 'worst imaginable pain').

CONTACTS AND LOCATIONS:
Overall Officials: Ayhan Sönmez, Study Director — SAMSUN UNİVERSİTY
Locations (1):
- Samsun training and research hospital, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No